CLINICAL TRIAL: NCT02976012
Title: Endolaserless Vitrectomy With Intravitreal Aflibercept Injection for Proliferative Diabetic Retinopathy-Related Vitreous Hemorrhage (LASER LESS TRIAL)
Brief Title: Endolaserless Vitrectomy With Intravitreal IAI for PDR-Related VH
Acronym: LASERLESS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast Retina Center, Georgia (Other)
Responsible Party: Principal Investigator, Dennis M. Marcus, M.D., Principal Investigator, Southeast Retina Center, Georgia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGFTe-DR-1548
Record Dates: First submitted 2015-11-04; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Proliferative Diabetic Retinopathy; Aflibercept; Vitreous Hemorrhage
MeSH Terms: conditions — Vitreous Hemorrhage | interventions — aflibercept; Intravitreal Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IAI q8 week Group (Active Comparator): Eyes will be randomized on the day of endolaserless vitrectomy surgery or first postoperative 1-2 week visit to a group ("q8 week Group") where 4 additional mandatory postoperative q4weeks IAI followed by mandatory q8 weeks IAI for 52 weeks follow-up. Starting at week 20 in the q8week group eyes may be eligible to receive additional 2mg IAI (intravitreal aflibercept) (monthly) treatment
  Interventions: Drug: Aflibercept; Procedure: Endolaserless Vitrectomy
- IAI q16 week Group (Active Comparator): Eyes will be randomized on the day of endolaserless vitrectomy surgery or first postoperative 1-2 week visit to a group (q16week Group) where 2 additional mandatory postoperative q4weeks IAI will be followed by mandatory q16weeks IAI for 52 weeks follow-up. Starting at week 12 in the q16 group, eyes may be eligible to receive additional 2mg IAI (intravitreal aflibercept) (monthly) treatment.
  Interventions: Drug: Aflibercept; Procedure: Endolaserless Vitrectomy

INTERVENTIONS:
Drug: Aflibercept — . Study eyes will receive one preoperative intravitreal aflibercept injection (IAI) <21 days prior to vitrectomy and one intraoperative intravitreal aflibercept at end of surgery. Eyes will be randomized on the day of surgery or 1-2 weeks post-operatively to either a q8week IAI dosing regimen group or a q16week IAI dosing regimen group.
  Other Names: Eylea; 2 mg/0.05 mL single use vial for intravitreal injection
Procedure: Endolaserless Vitrectomy — Endolaserless vitrectomy and intraoperative and postoperative IAI in patients with PDR-related vitreous hemorrhage

SUMMARY:
This is a phase I/II open label, randomized, interventional clinical trial. Study eyes will receive one preoperative intravitreal aflibercept injection (IAI) <21 days but >7 days prior to vitrectomy and one intraoperative IAI at end of surgery followed by randomization in a 1:1 ratio into either 4 mandatory postoperative q4weeks IAI followed by mandatory q8 weeks IAI for 52 weeks follow-up (q8 week Group) or 2 mandatory postoperative q4weeks IAI followed by mandatory q16 weeks IAI for 52 weeks follow-up (q16 week Group).

DETAILED DESCRIPTION:
This is a phase I/II open label, randomized, interventional clinical trial. Study eyes will receive one preoperative intravitreal aflibercept injection (IAI) <21 days but >7 days prior to vitrectomy and one intraoperative intravitreal aflibercept at end of surgery followed by randomization in a 1:1 ratio into either 4 mandatory postoperative q4weeks IAI followed by mandatory q8 weeks IAI for 52 weeks follow-up (q8 week Group) or 2 mandatory postoperative q4weeks IAI followed by mandatory q16 weeks IAI for 52 weeks follow-up (q16 week Group).

Follow-up visits occur 1 day and 1-2 weeks, and 4 weeks postoperatively and then every 4 weeks from the first postoperative IAI for 52 weeks. One preoperative visit and every postoperative visit (except day one postoperatively) will include ETDRS Best Corrected Visual Acuity (BCVA), Intraocular Pressure (IOP) measurement, Slit lamp biomicroscopy, Indirect ophthalmoscopy, Heidelberg Spectralis Spectral Domain Optical Coherence Tomography (SD-OCT) (no OCT for preoperative visit) and evaluation for systemic and ocular adverse events. Seven standard field photographs and Optos wide-field fluorescein angiography will be performed at postoperative visits at 4, 16, 28, 40,and 52 weeks. Humphrey visual field (HVF) testing (30-2 and 60-4 test patterns) will be performed at postoperative visits at 4 and 52 weeks. Preoperative B scan echography will be required standard of care(SOC) to assess for macular traction, non-macular traction, retinal detachment and vitreous hemorrhage(VH). Identification of traction macular detachment will exclude the patient from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age >18 years with Diabetes Mellitus
2. PDR- related vitreous hemorrhage and not of another cause
3. BCVA Vision LP or better
4. Investigator determination that vitrectomy indicated for PDR-related vitreous hemorrhage
5. Willing and able to comply with clinic visits and study-related procedures
6. Provide HIPPA and signed informed consent prior to any study procedures

Exclusion Criteria:

1. A condition per investigator opinion, would preclude participation in the study (unstable medical status, cardiovascular disease, glycemic control, inability to follow up etc.)
2. Participation in an investigational trial within 30 days of enrollment
3. Known allergy to IAI
4. Systemic anti-VEGF or pro-VEGF treatment within 4 months of enrollment
5. For women of childbearing age, pregnant or lactating or intending to become pregnant within the next 3 years
6. History of PRP or peripheral retinal cryopexy or peripheral retinopexy for any reason in the study eye
7. History of vitrectomy in the study eye
8. History or evidence for rhegmatogenous retinal detachment in the study eye
9. Evidence of traction retinal detachment involving or threatening central macula in the study eye
10. Exam evident of external ocular infection (i.e. conjunctivitis, significant blepharitis, chalazion etc)
11. Intravitreal anti-VEGF injection in the study eye <4weeks from enrollment.
12. Pregnant or breast-feeding women
13. Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly) *Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
• Ocular and systemic safety evaluation for adverse events at any time point through 52 weeks: | Through 52 weeks from Baseline
  Examples include worsened acuity >30 letters, rhegmatogenous or tractional retinal detachment, endophthalmitis, new or increased vitreous hemorrhage, cataract progression or surgery, need for additional vitrectomy or scleral buckle, development of new DME after OCT documentation of absence of DME, systemic thromboembolic events, deaths and systemic serious adverse events at any time point through week 52.

SECONDARY OUTCOMES:
Mean change in BCVA letter score | 52 weeks from Baseline
  Mean change in BCVA letter score over time through week 52
Mean BCVA letter score | 52 weeks from Baseline
  Mean BCVA letter score over time through week 52
Proportion of eyes with progression of PDR | Through 52 weeks from Baseline
  Proportion of eyes with progression of PDR as defined above at any time point through week 52
Mean OCT CSF thickness | Through 52 weeks from Baseline
  Mean OCT CSF thickness over time through week 52
Proportion of eyes with OCT CSF thickness <300um | Through 52 weeks from Baseline
  Proportion of eyes with OCT CSF thickness <300um at week 52
Proportion of eyes with absence of Optos widefield fluorescein angiographic macular leakage | Through 52 weeks from Baseline
  Proportion of eyes with absence of Optos widefield fluorescein angiographic macular leakage at week 52
Proportion of eyes with absence of active neovascularization | Through 52 weeks from Baseline
  Proportion of eyes with absence of active neovascularization by Optos widefield fluorescein angiography at week 52
Proportion of eyes with absence of active neovascularization | Through 52 weeks from Baseline
  Proportion of eyes with absence of active neovascularization by 7 standard field photography at week 52
Proportion of eyes with unchanged, worsened, or improved fluorescein angiographic macular leakage | Through 52 weeks from Baseline
  Proportion of eyes with unchanged, worsened, or improved fluorescein angiographic macular leakage from baseline angiograms at week 52
Proportion of eyes with unchanged, worsened, or improved fluorescein angiographic neovascularization | Through 52 weeks from Baseline
  Proportion of eyes with unchanged, worsened, or improved fluorescein angiographic neovascularization from baseline angiograms at week 52
Proportion of eyes with unchanged, worsened, or improved fundus photographic DME appearance | Through 52 weeks from Baseline
  Proportion of eyes with unchanged, worsened, or improved fundus photographic DME appearance from baseline photographs at week 52
Mean cumulative score and change for the combined 30-2 and 60-4 HVF test | Through 52 weeks from Baseline
  Mean cumulative score and change for the combined 30-2 and 60-4 HVF test from week 4 to week 52.
Proportion of eyes requiring additional IAI other than mandatory injections | Through 52 weeks from Baseline
  Proportion of eyes requiring additional IAI other than mandatory injections through week 52
Proportion of eye with progression of PDR requiring rescue PRP standard of care | Through 52 weeks from Baseline
  Proportion of eye with progression of PDR requiring rescue PRP standard of care at any time point through 52 weeks
Proportion of eyes requiring PRP or retinopexy | Through 52 weeks from Baseline
  Proportion of eyes requiring PRP or retinopexy through week 52
Proportion of eyes requiring additional vitrectomy | Through 52 weeks from Baseline
  Proportion of eyes requiring additional vitrectomy through week 52
Proportion of enrolled eyes requiring intraoperative endolaser in a PRP pattern at the time of initial vitrectomy | Through 52 weeks from Baseline
  Proportion of enrolled eyes requiring intraoperative endolaser in a PRP pattern at the time of initial vitrectomy

CONTACTS AND LOCATIONS:
Overall Officials: Dennis M Marcus, MD, Principal Investigator — Southeast Retina Center, PC
Locations (1):
- Southeast Retina Center, PC, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided